CLINICAL TRIAL: NCT07149935
Title: Continuous Effect Of Long-Term Rehabilitation Training On Clinical Improvement(TTCI) And Cardiopulmonary Function In Pulmonary Arterial Hypertension Patients- A Multicenter-randomisation Study
Brief Title: Continuous Effect Of Rehabilitation Training On Pulmonary Arterial Hypertension Patients
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: RenJi Hospital (Other)
Collaborators: Shanghai Pulmonary Hospital, Shanghai, China (Other); Shanghai General Hospital, Shanghai Jiao Tong University School of Medicine (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: Rehabilitation of PAH
Record Dates: First submitted 2024-06-05; First posted 2025-09-02 (Actual); Last update posted 2025-09-02 (Actual); Status verified 2025-08

CONDITIONS: Pulmonary Hypertension
Keywords: Rehabilitation, Pumonary arterial hypertension
MeSH Terms: conditions — Hypertension, Pulmonary

STUDY DESIGN:
Intervention Model Description: The recruited patients were divided into two groups after random allocation.
  Group C (control): this group was the control group, in which patients did not receive rehabilitation training; they only received targeted drug therapy, health education and daily activities.
  Group T (treatment): this group of subjects is the treatment group, in the treatment group, in addition to receiving targeted drug therapy, daily activities, but also under medical supervision to carry out appropriate rehabilitation training.
Masking Description: Because the specificity of rehabilization, it is not suitable for us to mask
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- rehabilitation training (Experimental): open label
  Interventions: Other: Rehabilitation Training
- control (No Intervention): open label

INTERVENTIONS:
Other: Rehabilitation Training — The rehabilitation training has two parts: the exercise training at home（5 times per week, as well as the Inspiratory muscle training(once per day) including Respiratory trainer exercise and abdominal breathing training.
  Arms: rehabilitation training

SUMMARY:
This multicenter, open label, double-arm study aims at investigating the the continuous effect of long-Term rehabilitation training on clinical improvement(ITTCI) and cardiopulmonary function in pulmonary arterial hypertension patients

DETAILED DESCRIPTION:
Pulmonary Arterial Hypertension (PAH) is a disease caused by various reasons leading to pulmonary vascular remodelling and then results in a progressive increase in pulmonary vascular resistance and right heart failure. PAH progresses rapidly,with a poor prognosis. Targeted drugs has brought about an improvement in the quality of life of patients with PAH. However, in most cases, patients' clinical symptoms will be gradually worsen with exercise capacity gradually declining. The prognosis of PAH remains bleak. Although exercise was previously considered as a relative contraindication for PAH patients , a growing body of research has found that exercise rehabilitation is safe and effective for them. Patients show greater improvement in their symptoms and quality of life. Effective and appropriate exercise rehabilitation in low- and middle-income countries can maximise the therapeutic benefits of targeted medication, improve patient survival rate, and enhance exercise tolerance and cardiorespiratory fitness. In this study, we will investigate the continuous effects of exercise rehabilitation on the clinical improvement (time to clinical improvement, TTCI) and cardiorespiratory fitness over a 1-year period of long-term rehabilitation, including aerobic training (aerobic power cycling and treadmill walking) and inspiratory muscle training (respiratory trainer and lip-contracting abdominal breathing).

ELIGIBILITY:
Inclusion Criteria:

1. Patients who suffered from pre-capillary PAH (mPAP ≥ 20 mmHg, PVR > 2 Woods unit, PAWP ≤ 15 mmHg) confirmed by right heart catheterisation.
2. Patients who are in the status of WHO-FC I-III.
3. Patients between 18 and 75 years old
4. Female subjects are not pregnant.
5. Patients are treated with PAH-targeted drugs and are in a stable state and there is no progress of disease).
6. Patients have not received exercise rehabilitation training within six months.

Exclusion Criteria:

Patients with the following diseases or symptoms:

1. Pulmonary vascular occlusive disease
2. Respiratory diseases
3. Ischaemic heart disease, complex congenital heart disease (e.g., tetralogy of Fallot, etc.), cardiomyopathy, valvular disease
4. Active liver disease
5. Severe kidney disease
6. Motor disorders (e.g. lower limb fracture, ataxia, etc.)
7. Malignant tumour diseases
8. Physical disability
9. Hb ≤ 80g / L
10. Systolic blood pressure ≤85mmHg
11. History of syncope within 3 months
12. History of supraventricular or ventricular arrhythmia at rest within 3 months.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 104 (Estimated)
Dates: Start 2024-09-01 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
6 minutes walk distance（ 6MWD） | every 3 months, until 6 months
  The walk distance of patients in 6 minutes
Improved Time To Clinical Improvement(ITTWI) | every 3 months, until 6months
  The time that required from the time of rehabilitation training to the first occurrence of at least one stratum improvement of the weber classification

SECONDARY OUTCOMES:
Echocardiographic index---right ventricle | every 3 months, until 6 months
  TAPSE, right ventricular diameter, tricuspid annular systolic motion s'
Echocardiographic index---left ventricle | every 3 months, until 6 months
  left intraventricular diameter, diastolic left ventricular eccentricity index, systolic left ventricular eccentricity index
Echocardiographic index---left ventricle | every 3 months, until 6months
  TAPSE/PASP
CPET index | every 3 months, until 6months
  AT, VE/VCO2 slope, PetCO2, oxygen pulse (VO2/HR), peak oxygen uptake (peak VO2),VE/VO2,PetO2
SF-36 score | every 3 months, until 6months
  SF-36 is a scale for evaluating the life quality of PAH patients
Echocardiographic index-others | every 3 months, until 6months
  RVFAC（right ventricle fraction of area changes）, diameter of pulmonary artery

CONTACTS AND LOCATIONS:
Overall Officials: Jieyan Shen, PhD, Study Chair — Shanghai Jiao Tong University School of Medicine Affiliated Renji Hospital
Locations (1):
- Renji Hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No